CLINICAL TRIAL: NCT04870697
Title: Effects of Acceptance and Commitment Therapy on Promoting Parental Quality of Life and Reducing Psychological Distress in Parents of Children With Cancer: A Randomized Controlled Trial Protocol
Brief Title: Acceptance and Commitment Therapy for Parents of Children With Cancer
Acronym: ACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Xiaohuan Jin, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CREC Ref. No 2020.452
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Childhood Cancer
Keywords: parents; Acceptance and Commitment Therapy; psychological flexibility; psychological distress; quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT group (Experimental): In addition to usual care, participants in the ACT group will receive ACT intervention. ACT intervention will be conducted in an individual-based format with four weekly sessions. The first session is a face-to-face format and the other three sessions are online live format.
  Interventions: Behavioral: ACT intervention
- Control group (Other): Participants in the control group will receive usual care in the study setting delivered by clinical staff. The rationale for adopting usual care as a control group is not only because it is more commonly used but also for practical and ethical considerations, as usual care is what is already being delivered clinically, therefore the results of the study can support any necessity of changes to clinical practice or not.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: ACT intervention — The components of ACT intervention will include six processes to foster parental PF according to the ACT framework.
  Session one - Generate creative hopelessness and build acceptance. The objective is to help parents know about the ACT intervention and realize the experiential avoidance or emotional control strategies do not work, finally turn attention to more useful strategies.
  Session two - Create space for your thought. The objective is to help parents create a distance from their thoughts and facilitate parents' ability of not being trapped by thoughts.
  Session three - Focus on here and now. The objectives to facilitate parents' experiences of observing self and contact with the present moment but not trapped in the past or future.
  Session four - Commit actions in line with the value. The objectives to help parents identify their inner value and take value-based actions even facing the challenges in current difficulties of their children with cancer.
  Arms: ACT group
Other: Usual care — Usual care in this study setting includes providing general information, education, psychological support, and consultation.
  Arms: Control group

SUMMARY:
The current study aims to develop a theoretically driven ACT intervention and examine its effects among parents of children with cancer. The objectives are:

1. To examine the effects of ACT intervention on parental QOL and psychological distress (symptoms of anxiety, depression and stress) in parents of children with cancer.
2. To examine the effects of ACT intervention on parental negative experience, experiential avoidance and psychological flexibility in parents of children with cancer.
3. To examine the effects of ACT intervention on psychological adjustment of children with cancer.

DETAILED DESCRIPTION:
A pilot study will be used to evaluate the feasibility and acceptability of ACT intervention protocol in Chinese parents of children with cancer. A two-arm parallel randomized controlled trial (RCT) will be used to evaluate the effects of ACT intervention in parents of children with cancer.

Eligible participants will be randomly assigned into a 1:1 allocation ratio to the ACT group or control group using block randomization with random mixture blocks of 4, 6 and 8. This can avoid the greater frequency of assignments to either group and lead to more balanced treatment groups in size and key outcome-related characteristics over time while reducing the predictability of assignment from the preceding assignment. A sequence list of two group labels (1 = ACT group, 2 = Control group) will be generated using a computerized generation randomization tool by an independent statistician who is blinded to the meaning of group labels will not involve the other part of the study. The group allocation assignment labels will be contained in opaque sealed envelopes and concealed to all researchers and participants involved in this study until the research investigator has completed the assessments of the participant and obtained written consent during the recruitment.

Considering the nature of the study, blinding of participants and ACT interventionists will be impossible. The research assistants involved in data collection and data entry as well as health routine care providers in the units of study hospital will be blinded to the group allocation.

To prevent possible contamination, the ACT intervention for parents in the ACT group will be conducted in a meeting room in the staff area which is geographically separate from the patient area. Besides, the participants are required not to show ACT intervention materials to, nor discuss the intervention contents with other parents in the unit.

ELIGIBILITY:
Inclusion Criteria:

The parents will be recruited if parent-child dyads fulfill the following eligibility criteria

Parents:

* Over the ages of 18 years old
* Fathers or mothers who are the primary caregivers (provide the largest amount of daily care) of Children with cancer
* Living together with the childhood cancer patients
* Can communicate in Chinese and follow the instructions of the study
* Can be accessible by telephone or by email

Children:

* Between the ages of 2 to 17 years old
* Newly diagnosed of cancer by a physician in the previous six months and currently receive treatment

Exclusion Criteria:

* Parents or their child who were currently participating in another cancer-related intervention study
* Parents or their children who are cognitive impaired
* Children in critical condition or palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in parental quality of life at one week after the intervention | Baseline and one week after the intervention
  PedsQL Parent HRQL Scale is adopted to assess parental quality of life. PedsQL Parent HRQL Scale consists of 20 items with 4 subscales of physical functioning, emotional functioning, social functioning, and cognitive functioning. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (almost always). Higher scores indicate higher quality of life.
  Change = (One week after the intervention score - baseline score)
Change from baseline in parental quality of life at three months after the intervention | Baseline and three months after the intervention
  PedsQL Parent HRQL Scale is adopted to assess parental quality of life. PedsQL Parent HRQL Scale consists of 20 items with 4 subscales of physical functioning, emotional functioning, social functioning, and cognitive functioning. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (almost always). Higher scores indicate higher quality of life.
  Change = (Three months after the intervention score - baseline score)
Change from baseline in parental distress at one week after the intervention | Baseline and one week after the intervention
  Depression Anxiety Stress Scales-21 is adopted to assess the level of depression, anxiety and stress in parents with 21 items and 3 subscales. Each item is rated on a 4-point Likert scale ranging from 0 (never) to 3 (always). Higher scores indicate more severe symptoms of depression, anxiety, or stress.
  Change = (One week after the intervention score - baseline score)
Change from baseline in parental distress at three months after the intervention | Baseline and three months after the intervention
  Depression Anxiety Stress Scales-21 is adopted to assess the level of depression, anxiety and stress in parents with 21 items and 3 subscales. Each item is rated on a 4-point Likert scale ranging from 0 (never) to 3 (always). Higher scores indicate more severe symptoms of depression, anxiety, or stress.
  Change = (Three months after the intervention score - baseline score)

SECONDARY OUTCOMES:
Change from baseline in parental psychological experience of child Illness at one week after the intervention | Baseline and one week after the intervention
  Parent Experience of Child Illness is adopted to assess parental psychological experience of their children with cancer. The scale consists of 25 items with 4 subscales of 'guilt and worry', 'unresolved sorrow and anger', 'long-term uncertainty' and 'emotional resources'. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (always). Higher scores indicate more difficulties in adjustment to their children with cancer.
  Change = (One week after the intervention score - baseline score)
Change from baseline in parental psychological experience of child Illness at three months after the intervention | Baseline and three months after the intervention
  Parent Experience of Child Illness is adopted to assess parental psychological experience of their children with cancer. The scale consists of 25 items with 4 subscales of 'guilt and worry', 'unresolved sorrow and anger', 'long-term uncertainty' and 'emotional resources'. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (always). Higher scores indicate more difficulties in adjustment to their children with cancer.
  Change = (Three months after the intervention score - baseline score)
Change from baseline in parental experiential avoidance at one week after the intervention | Baseline and one week after the intervention
  Acceptance and Action Questionnaire-II is adopted to assess experiential avoidance of parents. AAQ-II consists of 7 items. Each item is rated on a 7-point Likert scale ranging from 1 (never) to 7 (always). A higher score indicates great experiential avoidance.
  Change = (One week after the intervention score - baseline score)
Change from baseline in parental experiential avoidance at three months after the intervention | Baseline and three months after the intervention
  Acceptance and Action Questionnaire-II is adopted to assess experiential avoidance of parents. AAQ-II consists of 7 items. Each item is rated on a 7-point Likert scale ranging from 1 (never) to 7 (always). A higher score indicates great experiential avoidance.
  Change = (Three months after the intervention score - baseline score)
Change from baseline in parental psychological flexibility at one week after the intervention | Baseline and one week after the intervention
  Comprehensive assessment of Acceptance and Commitment Therapy processes is adopted to assess psychological flexibility of parents. CompACT consists of 23 items to measure three dyadic processes of ACT on 'acceptance and defusion', 'present moment awareness' and 'self as values and committed action'. Each item is rated on a 7-point Likert scale ranging from 0 (never) to 6 (always). Higher scores indicate a lower level of PF.
  Change = (One week after the intervention score - baseline score)
Change from baseline in parental psychological flexibility at three months after the intervention | Baseline and three months after the intervention
  Comprehensive assessment of Acceptance and Commitment Therapy processes is adopted to assess psychological flexibility of parents. CompACT consists of 23 items to measure three dyadic processes of ACT on 'acceptance and defusion', 'present moment awareness' and 'self as values and committed action'. Each item is rated on a 7-point Likert scale ranging from 0 (never) to 6 (always). Higher scores indicate a lower level of PF.
  Change = (Three months after the intervention score - baseline score)
Change from baseline in psychological adjustment of children with cancer one week after the intervention | Baseline and one week after the intervention
  Strengths and Difficulties Questionnaire is adopted to assess the psychological adjustment of children ages 2 to 17 years old. SDQ consists of 25 items to measure the emotional symptoms and behavioural problems of children. Each item is rated on a 3-point Likert scale ranging from 0 (not true) to 2 (certainly true). A higher score indicates poor psychological adjustment.
  Change = (One week after the intervention score - baseline score)
Change from baseline in psychological adjustment of children with cancer at three months after the intervention | Baseline and three months after the intervention
  Strengths and Difficulties Questionnaire is adopted to assess the psychological adjustment of children ages 2 to 17 years old. SDQ consists of 25 items to measure the emotional symptoms and behavioural problems of children. Each item is rated on a 3-point Likert scale ranging from 0 (not true) to 2 (certainly true). A higher score indicates poor psychological adjustment.
  Change = (Three months after the intervention score - baseline score)

CONTACTS AND LOCATIONS:
Overall Officials: Cho Lee Wong, PhD, Study Director — Chinese University of Hong Kong
Locations (1):
- Children's Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No